CLINICAL TRIAL: NCT02861729
Title: Clinical Outcomes of Zirconia-reinforced Lithium Silicate Partial Coverage Crowns Compared to Lithium Disilicate Partial Coverage Crowns: A Randomized Controlled Clinical Trial
Brief Title: Clinical Outcomes of Zirconia-reinforced Lithium Silicate Partial Coverage Crowns Compared to Lithium Disilicate Partial Coverage Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Sayed abdo Hassan Nassar, PHD student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-08-177
Record Dates: First submitted 2016-08-04; First posted 2016-08-10 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Partial Coverage Restoration
Keywords: Partial coverage restoration; Crown; Posterior teeth; All ceramic; Zirconia reinforced lithium silicate; Lithium disilicate; CAD/CAM
MeSH Terms: interventions — VITA Suprinity

STUDY DESIGN:
Intervention Model Description: split-mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprinity (Experimental): Vita Suprinity® (VITA Zahnfabrik H. Rauter GmbH & Co.KG- Germany) Zirconia reinforced lithium silicate PCRs
  Interventions: Other: Vita Suprinity
- e.max (Active Comparator): IPS-e.max® CAD (Ivoclar Vivadent AG, Schaan - Liechtenstein) lithium disilicate PCRs
  Interventions: Other: IPS e.max

INTERVENTIONS:
Other: Vita Suprinity — zirconia reinforced lithium silicate partial coverage restorations
  Arms: Suprinity
Other: IPS e.max — lithium disilicate partial coverage restorations
  Arms: e.max

SUMMARY:
The purpose of this randomized controlled clinical trial is to evaluate the clinical outcomes of Partial Coverage Restorations fabricated with zirconia-reinforced lithium silicate ceramic system compared to partial coverage restorations fabricated with lithium disilicate ceramic system.

DETAILED DESCRIPTION:
This study is constructed to assess in patients with carious vital posterior teeth whether the use of Vita Suprinity® (VITA Zahnfabrik H. Rauter GmbH & Co.KG- Germany) Zirconia reinforced lithium silicate partial coverage restorations will result in higher survival rates and better patient related outcome scores compared to IPS-e.max® CAD (Ivoclar Vivadent AG, Schaan - Liechtenstein) lithium disilicate partial coverage restorations.

ELIGIBILITY:
Inclusion Criteria:

* Participants:
* Good oral hygiene, papillary bleeding index (PBI) < 35%.
* Positive patient acceptance to participate in the trial.

Teeth:

* Carious class II or MOD lesions
* Vital upper or lower posterior teeth with no signs of irreversible pulpitis.
* Normal occlusion
* Single tooth restoration (no edentulous space that requires fixed prosthesis)

Exclusion Criteria:

* Participants
* Pregnancy.
* Disabilities.
* Systemic disease or severe medical complications.
* Bad oral hygiene
* Heavy smoking.
* Xerostomia.
* Lack of compliance.
* Evidence of severe bruxism, clenching, or temporomandibular disorders.

Teeth:

* Deep carious defects (close to pulp, less than 1 mm distance).
* Periapical pathology or signs of pulpal pathology.
* Tooth hypersensitivity.
* Rampant caries.
* Non-vital or endodontically treated teeth.
* Sever periodontal affection.
* Tooth mobility

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Survival rate | 12 month
  Absolute failure is defined by clinical unacceptable fracture and crack development which required a replacement of the entire restoration, and/or secondary caries as well as endodontic complications

SECONDARY OUTCOMES:
Restorations with Marginal gap as assessed visually by US public health service criteria | 12 month
  restorations with visually detectable margin, catch or penetration of explorer at baseline or a change from baseline on visual analogue scale at 12 month
Restorations with Marginal discoloration as assessed visually by US public health service criteria | 12 month
  restorations with visually detectable discoloration along margin at baseline or a change from baseline on visual analogue scale at 12 month
Restorations with color mismatch with adjacent teeth as assessed visually by US public health service criteria | 12 month
  restorations with visually detectable color mismatch with adjacent teeth at baseline or a change from baseline on visual analogue scale at 12 month
Restorations with surface roughness as assessed tactilely by US public health service criteria | 12 month
  restorations with tactilely detectable rough surface at baseline or a change from baseline on visual analogue scale at 12 month
Restorations developed secondary caries as assessed visually by US public health service criteria | 12 month
  restorations with visually detectable secondary caries at baseline or a change from baseline on visual analogue scale at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Katamish, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guess PC, Strub JR, Steinhart N, Wolkewitz M, Stappert CF. All-ceramic partial coverage restorations--midterm results of a 5-year prospective clinical splitmouth study. J Dent. 2009 Aug;37(8):627-37. doi: 10.1016/j.jdent.2009.04.006. Epub 2009 May 3. PMID 19477570
- [Background] Stappert CF, Guess PC, Chitmongkolsuk S, Gerds T, Strub JR. All-ceramic partial coverage restorations on natural molars. Masticatory fatigue loading and fracture resistance. Am J Dent. 2007 Feb;20(1):21-6. PMID 17380803
- [Background] Guess PC, Stappert CF. Midterm results of a 5-year prospective clinical investigation of extended ceramic veneers. Dent Mater. 2008 Jun;24(6):804-13. doi: 10.1016/j.dental.2007.09.009. Epub 2007 Nov 19. PMID 18006051
- [Background] Rinke S, Pabel AK, Rodiger M, Ziebolz D. Chairside Fabrication of an All-Ceramic Partial Crown Using a Zirconia-Reinforced Lithium Silicate Ceramic. Case Rep Dent. 2016;2016:1354186. doi: 10.1155/2016/1354186. Epub 2016 Mar 6. PMID 27042362
- [Background] McDonald A. Preparation guidelines for full and partial coverage ceramic restorations. Dent Update. 2001 Mar;28(2):84-90. doi: 10.12968/denu.2001.28.2.84. PMID 11819962
- [Background] Signore A, Benedicenti S, Covani U, Ravera G. A 4- to 6-year retrospective clinical study of cracked teeth restored with bonded indirect resin composite onlays. Int J Prosthodont. 2007 Nov-Dec;20(6):609-16. PMID 18069370
- [Background] Edelhoff D, Sorensen JA. Tooth structure removal associated with various preparation designs for posterior teeth. Int J Periodontics Restorative Dent. 2002 Jun;22(3):241-9. PMID 12186346
- [Background] Stappert CF, Chitmongkolsuk S, Silva NR, Att W, Strub JR. Effect of mouth-motion fatigue and thermal cycling on the marginal accuracy of partial coverage restorations made of various dental materials. Dent Mater. 2008 Sep;24(9):1248-57. doi: 10.1016/j.dental.2008.02.005. Epub 2008 Apr 18. PMID 18395785
- [Background] Murgueitio R, Bernal G. Three-year clinical follow-up of posterior teeth restored with leucite-reinforced ips empress onlays and partial veneer crowns. J Prosthodont. 2012 Jul;21(5):340-5. doi: 10.1111/j.1532-849X.2011.00837.x. Epub 2012 Feb 28. PMID 22372380
- [Background] Kois DE, Isvilanonda V, Chaiyabutr Y, Kois JC. Evaluation of fracture resistance and failure risks of posterior partial coverage restorations. J Esthet Restor Dent. 2013 Apr;25(2):110-22. doi: 10.1111/jerd.12018. Epub 2013 Mar 19. PMID 23617385
- [Background] Vogl V, Hiller KA, Buchalla W, Federlin M, Schmalz G. Controlled, prospective, randomized, clinical split-mouth evaluation of partial ceramic crowns luted with a new, universal adhesive system/resin cement: results after 18 months. Clin Oral Investig. 2016 Dec;20(9):2481-2492. doi: 10.1007/s00784-016-1779-2. Epub 2016 Mar 12. PMID 26971352